CLINICAL TRIAL: NCT04428515
Title: Pilot Study to Evaluate Photoacoustic Imaging in Head and Neck Cancer
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Senior Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 135-2018
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer
Keywords: Photoacoustic; Head and Neck; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiotherapy Response Monitoring: Those undergoing radiation therapy treatment to their lymph nodes upon diagnosis of head and neck cancer
  Interventions: Device: Photoacoustic Imaging System

INTERVENTIONS:
Device: Photoacoustic Imaging System — Photoacoustic Imaging investigate changes of measured PA markers and compare these to radiological assessment of response of lymph node involvement to chemoradiation therapy for head and neck cancer

SUMMARY:
In this study, PA imaging will be used to examine the physiological and physical changes in lymph node involvements of head and neck cancer during radiotherapy with or without chemotherapy. Our objective in this pilot study will be to evaluate if PA parameters change within the lymph node involvements during chemoradiation therapy over time. Our hope is to use this information to correlate the changes in measured PA parameters with radiological response.

DETAILED DESCRIPTION:
A trained clinical research coordinator will evaluate and authorize that each screened volunteer is a suitable subject for the study prior to enrolment. Written informed consent will be obtained from each participant prior to any clinical research scans to be performed on the subject. Those subjects who qualify will have their lymph node imaged using a PA imaging system. Up to 50 subjects will be recruited for this study.

Participants will be imaged 5 times over the course of radiotherapy regimen, which span up to 7 weeks. The patients will be assessed with MRI 10 to 12 weeks after the completion of Chemoradiation therapy as per the institution's standard of care. The lymph nodes will be measured by a staff radiologist, and the sizing information will be used to categorize patients into responders or non-responders. This information will be accessed using the patient's electronic medical record. Each patient will be assigned an anonymized accession number to the study that withholds any identifiers. There will be a complete accounting of all missing and excluded data, if any.

Although we do not anticipate any adverse events, all AEs will be documented in the CRF, and will be immediately reported to the REB, the overseeing physician responsible for the patient's care, and the study principal investigators.

Descriptive statistics (arithmetic mean, standard deviation, and coefficient of variation) and tabulation (stem and leaf plots) of study endpoints (absolute values and absolute value/comparator differences) will be used. PA datasets will be tested for normality, using a Shapiro-Wilk test (alpha=0.05). Comparative tests will use an independent t-test (or Mann Whitney test for normality violations) to compare the PA measurements between different breast masses (fibroadenomas, cysts, tumors).

In determining chemoradiation therapy evaluation, the primary endpoint, multiple linear regression models to relate study endpoints to subject characteristics and a logistic regression model will be used to build for multiparametric analysis of multiple PA parameters as a predictive model to pathological response. Descriptive statistics (frequency per scan, frequency per subject) and tabulation will be used to analyze the frequency of system malfunction.

Overall Survival Evaluation, the secondary endpoint, will use linear discriminant analysis to test for sensitivity, specificity and accuracy of the PA parameters as a diagnostic test. Receiver-operating characteristic will be used to test for PA cutoff values and a logistic regression model will be used to build for multiparametric analysis of multiple PA parameters as a predictive model to pathological response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed head and neck carcinoma which has not been treated with any first-line therapy and will be treated with radiotherapy
* Measurable disease by ultrasound, or MRI performed within 28 days prior to treatment
* Eastern Co-operative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 6 months
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to dosing:

  1. hemoglobin >90 mg/dL
  2. leukocytes >3,000/mL
  3. absolute neutrophil count >1,500/mL
  4. platelets >100,000/mL
  5. total bilirubin within normal institutional limits
  6. AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  7. creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional upper limit of normal
* Subjects must give appropriate written informed consent prior to participation in the study;
* Subjects must be able and willing to comply with the safety procedures during the Scanning Period;

Exclusion Criteria:

* Chemotherapy, radiotherapy, or major surgery within 4 weeks prior to registering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to registration
* Receiving any other investigational agents
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition
* Contraindications to radiotherapy such as but not limited to:

  1. previous radiotherapy to an involved area
  2. active collagen vascular disease
  3. genetic diseases associated with hyper-radiosensitivity
* Any clinically serious infections requiring systemic anti-bacterial, antifungal or antiviral therapy
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection,
* Symptomatic congestive heart failure, unstable angina pectoris, and cardiac arrhythmia
* History of active ongoing seizure disorder
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men or women with confirmed head and neck carcinoma and will be treated with radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2027-04-23 (Estimated)

PRIMARY OUTCOMES:
Correlation of response to treatment between photoacoustic parameters and final radiological outcome. measures of outcome. | 3 months
  The primary study endpoint will investigate changes of measured PA markers and compare these to radiological assessment of response of lymph node involvement to chemoradiation therapy for head and neck cancer. Changes in PA parameters will be made to a pre-treatment point over the course of treatment.

SECONDARY OUTCOMES:
Correlation between photoacoustic parameters and five-year overall survival. | 5 years
  The secondary study endpoint will correlate changes of measured PA markers to five-year overall survival (OS) of the same patient cohort. The survival status and of the patient cohort will be tracked after the treatment for five years based on the patient information system and follow up surveys if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Czarnota, PhD, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No